CLINICAL TRIAL: NCT01978002
Title: Sensory Sensitivity and Urinary Symptoms in the Female Population
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, James Clemens, Principal Investigator, University of Michigan
Other Study IDs: HUM00054279
Record Dates: First submitted 2013-10-25; First posted 2013-11-07 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Bladder Pain and Discomfort; Urinary Urgency and Frequency; Bothersome Symptoms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1 (Clinic Patients): Women who have documented urinary status from surveys completed.
  Interventions: Behavioral: Pain sensitivity testing
- Group 2 (Community Sample): Women who have a clinical diagnosis of IC/BPS or OAB, and who have undergone urodynamic testing within the preceding 6 months as part of their routine clinical care.
  Interventions: Behavioral: Pain sensitivity testing; Behavioral: Urodynamic testing

INTERVENTIONS:
Behavioral: Pain sensitivity testing
Behavioral: Urodynamic testing
  Groups: Group 2 (Community Sample)

SUMMARY:
Bladder pain and discomfort, as well as urinary urgency and frequency, are bothersome symptoms seen frequently in the general population. Clinical diagnostic terms used to describe these symptoms include interstitial cystitis (IC), bladder pain syndrome (BPS), chronic prostatitis, and overactive bladder (OAB), but there is tremendous overlap between these entities, and the distinction between them is based more on eminence than evidence.

Pain and/or sensory sensitivity has been suspected to play a role in the pathogenesis of both bladder pain and urinary urgency/frequency. However, no previous studies have investigated whether entities such as IC/BPS and OAB might merely represent different points in a continuum of bladder sensory sensitivity. Moreover, we know of no studies that have directly compared sensory sensitivity in the bladder to global (i.e. CNS-mediated) sensory sensitivity.

In the study, a team of investigators with complementary expertise will perform a population-based study assessing bladder and overall sensory sensitivity, in a cohort of women representative of the population with respect to the entire continuum of bladder pain (from none to severe), and symptoms of urgency/frequency. These individuals will undergo urodynamics to measure sensory sensitivity in the bladder, as well as pressure pain and auditory loudness thresholds. The Specific Aims are to demonstrate: 1) sensory sensitivity in the bladder is related to sensory sensitivity elsewhere in the body, suggesting a CNS-driven mechanism, and 2) individuals in the population with greater global sensory sensitivity will display: a) more bladder pain, b) more urgency/frequency, and c) other symptoms of centrally-mediated pain states, such as pain in regions other than the bladder, fatigue, and insomnia.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old

Exclusion Criteria:

* 1) Neurological disease or disorder affecting the bladder; 2) Previous augmentation cystoplasty or cystectomy; 3) Systemic autoimmune disorder (such as Crohn's Disease or Ulcerative Colitis, Lupus, Rheumatoid Arthritis; 4)History of pelvic cancer (colon, bladder, uterus, ovary); 5) Current major psychiatric disorder or other psychiatric or medical issues that would interfere with study participation (e.g. dementia, psychosis, upcoming major surgery, etc); 6) Current pregnancy. These exclusion criteria will be assessed at the time of the initial telephone interview.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 will be women with a clinical diagnosis of IC/BPS or OAB, at least 18 years of age, who have had urodynamic testing performed within the preceding 6 months. All of these subjects will complete the questionnaires, mechanical sensitivity testing, and auditory sensitivity testing
  Group 2 will be women recruited from the community sample, at least 18 years of age. All of these subjects will complete the questionnaires, mechanical sensitivity testing, and auditory sensitivity testing. Half of the subjects (n=30) will also undergo urodynamic testing to measure bladder sensitivity.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Urodynamics | 1 year
  Sensation, desire to void, strong desire to void, and maximum cystometric capacity
Auditory Sensory Sensitivity | 1 year
  Sensitivity for loudness threshold will be performed using pure tone acoustic stimuli at an octave frequency of 2000 Hz and signal range from 40 to 100 dB

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States